CLINICAL TRIAL: NCT06060119
Title: Comparison of Microneedling With Subepithelial Connective Tissue Auto Graft for Gingival Augmentation- A Randomized Case Control Trial
Brief Title: Comparison of Microneedling and CTG for Gingival Augmentation- A RCT
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Krishnadevaraya College of Dental Sciences & Hospital (Other)
Responsible Party: Principal Investigator, Dr Prabhuji MLV, HOD OF PERIODONTOLOGY, Krishnadevaraya College of Dental Sciences & Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KCDSHEC/IP/2022/S21
Record Dates: First submitted 2023-09-13; First posted 2023-09-29 (Actual); Last update posted 2023-09-29 (Actual); Status verified 2023-09

CONDITIONS: Gingival Phenotype
MeSH Terms: interventions — Percutaneous Collagen Induction

STUDY DESIGN:
Intervention Model Description: SAMPLING TECHNIQUE Purposive Sampling technique will be done. All the patients meeting the criteria will be screened and then 12 patients will be randomly allotted into either of the two groups. The treatment allocation to the test and control group will be assigned by means of a sealed envelope containing a code derived from a computer generated randomized list to receive either -
  1. TEST GROUP (n = 12) - Microneedling on the selected area.
  2. CONTROL GROUP (n = 12) - Subepithelial connective tissue grafting at the contralateral site
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Comparison of Microneedling for Gingival Augmentation- A Randomized Case Control Trial (Experimental): 1. TEST GROUP (n = 12) - Microneedling on the selected a non-steroidal anti-inflammatory drug (Tab Ibuprofen 400mg) and antibiotic Amoxicillin 500mg thrice daily for three days after meals will be prescribed. In patients allergic to Amoxicillin, Clindamycin 300mg thrice daily is prescribed13
  Interventions: Device: microneedling
- Comparison of Microneedling with for Gingival Augmentation- A Randomized Case Control Trial (Experimental): 2.CONTROL GROUP (n = 12) - Subepithelial connective tissue grafting at the contralateral site non-steroidal anti-inflammatory drug (Tab Ibuprofen 400mg) and antibiotic Amoxicillin 500mg thrice daily for three days after meals will be prescribed. In patients allergic to Amoxicillin, Clindamycin 300mg thrice daily is prescribed13
  Interventions: Device: microneedling

INTERVENTIONS:
Device: microneedling — The operative sites will be anaesthetized with 2% lignocaine hydrochloride with adrenaline(1:80,000).Electric microneedling pen device model THAPPINKTM is used. Microneedling is carried out on the isolated site involving one tooth mesially and distally and 1.5mm apical to marginal gingiva each for 30-40 second intermittently. When pin point bleeding observed on the area of gingiva it is irrigated with sterile saline solution. Patient will be instructed to refrain from consuming hot beverage and brushing in that area for one day to avoid mechanical trauma. A total of 4 session of micro needling procedure will be carried out in one subject at 10 days intervals upto 40days
  Other Names: Derma pen

SUMMARY:
The presence study is toComparison of Microneedling with Subepithelial Connective Tissue Auto Graft for Gingival Augmentation- A Randomized Case Control Trial. The trial is in accordance with the Consolidated Standards of Reporting Trials (CONSORT) criteria, 2010.

DETAILED DESCRIPTION:
The periodontal phenotype previously called as biotype is a reflection of gingiva and buccal bone thickness. It is a vital clinical parameter as it will determine whether there will be recession , dehiscence and fenestration or pocket formation.1Basically gingival epithelium provides a physical barrier to infection and protects the deeper structures thus, the gingival phenotype has major impact on the outcome of the restorative, regenerative, implant and orthodontic therapy.2 Common causes of recession are faulty toothbrushing ,tooth malposition, abnormal frenum attachment, trauma from occlusion and orthodontic tooth movement in labial direction.2 Gingiva can be classified as thick > 1mm and thin < 1mm according to recent 2017 world work shop classification.3 Traditionally, gingival augmentation is achieved using free gingival graft, connective tissue graft, soft tissue substitutes. Subepithelial connective tissue auto graft is still the gold standard. All of these technique's are invasive, complicated, technique senstive and do not have cost efficiency4, thus there is an on going reasearch for a more simpler non invasive method to increase gingival thickness.

Microneedling also knows as "percutaneous collagen induction therapy" is a novel and innovative method to thicken gingiva.5It involves creating several microinjuries in the form of inducing superficial bleeding points there by inducing a wound healing cascade which releases a few key soft tissue growth factor's such as platelet-derived growth factors, transforming growth factors, connective tissue growth factor and fibroblast growth factors.1 Fernandes has developed a percutaneous technology based on principals of microneedling to initiate natural post traumatic inflammatory reaction by using microneedles.6 The growthfactor's thus released post injury stimulate proliferation of new cells and transformation of fibroblast into collagen and elastin fiber, starting from 5th day up to 8th week. Newly formed fibers thicken the tissue during the process known as neocollagenesis. Fibroblasts also trigger neoangiogenesis by accelerating the proliferation of endothelial cells in the blood vessels. The tissue remodeling changes continue from 8 weeks up to 1 year.7 Thus, this non-invasive technique of microneedling will be compared to the time tested subepithelial connective tissue autograft to obtain a deeper insight over its feasibility.

ELIGIBILITY:
Inclusion Criteria:

* Patients > 18 years of age.
* Patients with esthetic concern .
* Patient under going orthodontic, prosthodontic, restorative treatment where thick gingiva is necessary.
* Systemically healthy subjects
* Full mouth plaque index,full mouth bleeding on probing score < or = 15
* Patient with palatal mucosa greater than 4mm

Exclusion Criteria:

* Previous periodontal surgery
* Patients with history of coagulation disorder
* Smoking habit
* Pregnant and lactating females
* Use of any

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Estimated)
Dates: Start 2023-11-28 (Estimated); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-07-30 (Estimated)

PRIMARY OUTCOMES:
OBJECTIVES OF THE STUDY: The primary outcomes measured will be : 1) Increase in gingival augmentation with microneedling | 6 months
  1. Increase in gingival augmentation with microneedling will be measured in (mm)
  2. Comparison of microneedling with subepithelial connective tissue graft for gingival thickness in(mm) digital calliper and spreader file

SECONDARY OUTCOMES:
thickness in mm | 6 months
  Increase KTW (keratinization tissue width) will be checked in digital calliper and spreader file

IPD SHARING:
Plan to Share IPD: No